CLINICAL TRIAL: NCT02976896
Title: Efficacy and Safety of Apatinib Mesylate in Recurrent/Metastatic Esophageal Squamous Cell Carcinoma After the Failure of Conventional Treatment: a Phase II Clinical Trial
Brief Title: Apatinib for Esophageal Squamous Cell Cancer After the Failure of Standard Treatment
Acronym: Poetry-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhong Li (Other)
Responsible Party: Sponsor-Investigator, Yuhong Li, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Poetry-1
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apatinib Mesylate (Experimental): Patients will receive Apatinib Mesylate at 500mg/times,oral one times daily for 28 days.
  Interventions: Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Apatinib Mesylate — Patients will receive Apatinib Mesylate at 500mg/times,oral one times daily for 28 days.

SUMMARY:
We conduct the phase II clinical trial to further explore the efficacy and safety of Apatinib Mesylate in treating recurrent or metastatic esophageal squamous cell carcinoma after the failure of conventional treatments. An exploratory molecular marker analysis will be performed in order to find out the beneficial population of Apatinib Mesylate.

DETAILED DESCRIPTION:
Esophageal cancer is one of the most common malignant tumor in China. In Asian countries, esophageal squamous cell carcinoma is the main pathological type of esophageal carcinoma. Prognosis of esophageal squamous cell carcinoma is usually poor and surgery is the only radical treatment. Cisplatin (DDP, cisplatin), 5 - Fluorouracil (5 - Fluorouracil, 5 - FU) and taxane are the most adopted chemotherapy agents, with efficacy rates of 33%-40% as first-line treatment for metastatic or recurrent esophageal squamous carcinoma and a median overall survival of 6-10 months. New agents were needed. Apatinib Mesylate is a small molecule VEGFR tyrosine kinase inhibitor. The anti-tumor mechanism of Apatinib is inhibiting angiogenesis in malignancy by inhibiting VEGFR. Apatinib Mesylate was approved by CFDA (China Food and Drug Administration) for the treatment of advanced gastric cancer. In the previous clinical practice, we observed that part of the patients with esophageal squamous cell carcinoma were resistant to conventional treatments benefited from Apatinib Mesylate. Based on the research situation mentioned above, we decided to conduct a phase II clinical trial to further explore the efficacy and safety of Apatinib Mesylate in treating recurrent or metastatic esophageal squamous cell carcinoma after the failure of conventional treatments. An exploratory molecular marker analysis will be performed in order to find out the beneficial population of Apatinib Mesylate.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, age:18-75 years old.
2. The ECOG physical status score: 0 to 2.
3. Confirmed by histology of recurrent or metastatic esophageal squamous cell carcinoma.
4. Patients who previously received at least fluorouracil, platin or taxane-based palliative chemotherapy but failed(including patients who developed disease progression within half of a year after finishing their adjuvant or neoadjuvant chemotherapy) and patients who are intolerable or refuse to receive chemotherapy of agents mentioned above and develop disease progression within 2 months.
5. Never received treatment of apatinib or any other anti-angiogenesis agent, such as sorafenib, sunitinib, bevacizumab, endostar etc.
6. Lesions can be measured at single diameter by thoracic or abdominal computed tomography (CT) or magnetic resonance (MRI).Conventional methods should set at least 20mm as diameter or spiral CT 10 mm. Patients with increased or new lesions in radiotherapy area can be enrolled in the trial.
7. Expected survival ≥ 3 months.
8. If the subject have received surgery, the operative wound should be completely healed and without bleeding tendency.
9. Baseline of blood routine and biochemical routine should meet the following criteria:

   * ANC≥1.5×10^9/L（1500/mm3）
   * PLT≥75×10^9/L
   * Hb≥9 g/dL
   * Serum bilirubin levels no higher than 2 times the upper limit of normal value.
   * AST and ALT no higher than 2.5 times the upper limit of normal value(no higher than 5 times the upper limit of normal value when patients developed liver metastasis).
   * Serum creatinine no higher than 1.5 times the upper limit of normal value.
10. No malabsorption or other gastrointestinal disorders that will affect drugs absorption.
11. No severe complications such as active digestive tract hemorrhage, perforation, jaundice, gastrointestinal obstruction, non-cancerous fever > 38 ℃.
12. Patients should be voluntary to the trial and provide with signed informed consent.
13. Patients should have good compliance and cooperate with the evaluation of efficacy and adverse events and follow-ups according to the research plan.

Exclusion Criteria:

1. Evidence of gastrointestinal bleeding tendency including: local active ulcer lesions with occult blood (+ +); melena and haematemesis within 2 months; possibilities of digestive tract hemorrhage.
2. Evidence of hypertension that could not be controlled by drugs (SBP>140 mmHg, DBP>90 mmHg), grade I coronary heart disease, grade I arrhythmia(including QT interval prolonged by 450ms in male and 470ms in female) and grade I heart failure.
3. Evidence of severe postoperative complications including intestinal obstruction, anastomotic fistula, pancreatic fistula and anastomotic stenosis.
4. Evidence of urine protein ≥ (++) and 24 hours urinary protein quantitation >1.0 g.
5. Fractures unhealed for long term or incompletely healed.
6. Evidence of immunodeficiency disease, or other acquired or congenital immunodeficiency disease, or organ transplantation.
7. Evidence of coagulation disorders (INR>1.5, APTT>1.5 ULN), bleeding tendency(INR should be in normal value without anticoagulation 14 days before randomization), usage of anticoagulation or Vit K antagonist including warfarin, heparin or any other analogue. When INR≤ 1.5, small dosage of warfarin(1 mg p.o, qd) or Aspirin (dosage < 100mg/d) in preventive purpose is allowed.
8. Evidence of arterial/venous thrombotic events within 1 year before inclusion, including cerebrovascular accident (including TIA), deep vein thrombosis( vein thrombosis caused by venous catheterization in previous chemotherapy is excluded) and pulmonary embolism.
9. Known severe hypersensitivity to Apatinib or any of the excipients of this product
10. Severe systemic disease out of control such as unstable or uncompensated respiratory,cardiac,liver,renal diseases.
11. CNS metastases without radiotherapy and/or surgery. Patients with treated CNS metastases may participate in this trial,except for those who must receive hormone therapy and those whose prior hormone therapy for CNS metastases is less than 4 weeks.
12. psychiatric illness that would prevent the patient from giving informed consent
13. Patient has a concurrent malignancy or has a malignancy within 5 years of study enrollment, with the exception of nonmelanoma skin cancer or cervical carcinoma in situ
14. Patient is concurrently using other approved or investigational antineoplastic agent
15. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Disease control rate | 6 months

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Time to progression | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Incidence of Treatment-Emergent Adverse Events | Each follow up vist, assessed up to 12 months
  Safety evaluation according to the CTCAE4.0 standard, once every 1 cycle assessment
Quality of life using EORTC QLQ C30 - scale | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Life quality evaluation using EORTC QLQ C30 - scale，once every 1 cycle assessment
Quality of life using esophageal special scale QLQ - OES18 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Life quality evaluation using esophageal special scale QLQ - OES18, once every 1 cycle assessment

CONTACTS AND LOCATIONS:
Overall Officials: Li Yuhong, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes